CLINICAL TRIAL: NCT03764748
Title: Efficacy and Safety of Washed Microbiota Transplantation for Tourette's Syndrome
Brief Title: Washed Microbiota Transplantation for Tourette's Syndrome
Acronym: WMT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WMT-TS
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Tourette Syndrome
Keywords: Tic Disorders; Gut microbiota; Brain-gut axis; Washed Microbiota Transplantation; Tourette syndrome
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Washed microbiota transplantation (Experimental): WMT
  Interventions: Drug: Washed Microbiota Transplantation

INTERVENTIONS:
Drug: Washed Microbiota Transplantation — The prepared microbiota suspension was infused into the participates' lower gut.
  Other Names: Fecal microbiota transplantation

SUMMARY:
This study aimed to evaluate the efficacy of washed microbiota transplantation in the treatment of Tourette's syndrome (TS).

DETAILED DESCRIPTION:
Emerging scientific data support the significant role of microbiota in the modulation of the central nervous system. The reconstitution of gut microbiota might be a potential option to treat Tourette's syndrome (TS). FMT has been reported to be a highly effective therapy to restore the gut microbiota dysbiosis by transferring gut microbiota from healthy donors to patients. The newly improved methodology of FMT based on the automatic washing process and the related delivering consideration was named as washed microbiota transplantation (WMT) by the FMT-standardization study group. FMT has shown treatment potential in several gut-brain axis-related disorders, such as amyotrophic lateral sclerosis and Parkinson's disease, promoting us to investigate its treatment potential for Tourette's syndrome. In this study, investigators aimed to evaluate the efficacy of WMT for Tourette's syndrome and its comorbidities using specialized questionnaires for Tourette's syndrome and investigate the underlying mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were aged 6 to 17 years (inclusive);
2. Met the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria for TS;
3. Had a Yale Global Tic Severity Scale-Total Tic Score (YGTSS-TTS) of at least 20 at screening and baseline.
4. Underwent WMT.

Exclusion Criteria:

1. Complicated with certain brain disease, including tumor,injury,cerebrovascular disease;
2. Complicated with other severe disease, including cancers, organ failure, heart diseases;
3. Stereotypy associated with autism spectrum disorder;
4. With a confirmed diagnosis of psychiatric diseases, such as bipolar disorders; schizophrenia and major depressive disorders;
5. Clinically significant obsessive-compulsive disorder at baseline considered to be the primary cause of impairment at baseline;
6. Medications use affecting gut microbiota such as antibiotics and probiotics three months before WMT.
7. Other neurologic disorders other than TS that could influence the evaluation of tics.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
The change of Yale Global Tic Severity Scale-Total Tic Score (YGTSS-TTS) | baseline, 4 weeks, 8 weeks, 12 weeks, 6 months post transplantation
  The YGTSS rating scale is a semistructured clinician- or investigator-administered rating instrument in which participants or caregivers evaluate the number, frequency, intensity, complexity, and interference of motor and phonic tics in the prior week on a 6-point scale from 0 (none) to 5 (severe) [1]. The total Motor Tic Severity Score (MTSS; 0-25 points) is added to the total Vocal Tic Severity Score (VTSS; 0-25 points) to determine the TTS (0-50 points).

SECONDARY OUTCOMES:
the Clinical Global Impressions-Improvement scale | 4 weeks, 8 weeks, 12 weeks, 6 months post transplantation
  Positive treatment response was defined by a score of 1 (very much improved) or 2 (much improved) on the Clinical Global Impressions-Improvement scale. The Clinical Global Impression - Improvement scale is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as:1.Very much improved; 2.Much improved; 3. Minimally improved; 4. No change; 5. Minimally worse; 6. Much worse; 7.Very much worse.
the change of Gilles de la Tourette Syndrome Quality-of-Life Scale score | baseline, 4 weeks, 8 weeks, 12 weeks, 6 months post transplantation
  The Gilles de la Tourette Syndrome Quality-of-Life Scale with 27 items addresses the issue of how the illness affects patients' well-being. It ranges from 0 to108, and higher values represent a worse outcome.
the change of The Swanson, Nolan, and Pelham IV Scale (SNAP-IV) | baseline, 4 weeks, 8 weeks, 12 weeks, 6 months post transplantation
  It is an 26-item questionnaire that measured three of the ADHD symptoms, inattention, hyperactivity and oppositional defiant disorder. The 26-item checklist is scored on a 4-point Likert scale ranging between Not At All (0) and Very Much (3).
change of the Sleep Disturbance Scale for Children (SDSC) | baseline, 4 weeks, 8 weeks, 12 weeks, 6 months post transplantation
  The SDSC was 26-item test measuring sleep problems and each item received a value from 0 to 4, with higher scores indicating more severe sleep disorders.
change of the Gastrointestinal Symptom Rating Scale (GSRS) . | baseline, 4 weeks, 8 weeks, 12 weeks, 6 months post transplantation
  It is based on 15 questions which are scored into 5 domains: abdominal pain, reﬂux, indigestion, diarrhea, and constipation. Each item weights from 1 to 7, with higher scores reflecting more severe symptoms.
the difference of the gut microbe composition between individuals with TS and healthy children by sequencing faecal metagenome. | baseline, 12 weeks, 6 months post transplantation
  The composition of the gut microbiota is evaluated by sequencing faecal metagenome. We evaluate the differences in the structure of the flora and its metabolism between individuals with TS and control children at the phylum, genus and species levels of the intestinal flora, and to develop a model for predicting the structure of the flora.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD; PHD, Study Chair — The Second Hospital of Nanjing Medical University
Locations (2):
- China (2):
  - Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - SIR RUN RUN hospital of Nanjing Medical University, Nanjing, Jiangsu

REFERENCES:
- [Background] Hoffman BU, Lumpkin EA. A gut feeling. Science. 2018 Sep 21;361(6408):1203-1204. doi: 10.1126/science.aau9973. No abstract available. PMID 30237346
- [Background] Foster JA. Targeting the Microbiome for Mental Health: Hype or Hope? Biol Psychiatry. 2017 Oct 1;82(7):456-457. doi: 10.1016/j.biopsych.2017.08.002. No abstract available. PMID 28870296
- [Background] Roessner V, Plessen KJ, Rothenberger A, Ludolph AG, Rizzo R, Skov L, Strand G, Stern JS, Termine C, Hoekstra PJ; ESSTS Guidelines Group. European clinical guidelines for Tourette syndrome and other tic disorders. Part II: pharmacological treatment. Eur Child Adolesc Psychiatry. 2011 Apr;20(4):173-96. doi: 10.1007/s00787-011-0163-7. PMID 21445724
- [Background] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065
- [Background] Zhang F, Cui B, He X, Nie Y, Wu K, Fan D; FMT-standardization Study Group. Microbiota transplantation: concept, methodology and strategy for its modernization. Protein Cell. 2018 May;9(5):462-473. doi: 10.1007/s13238-018-0541-8. Epub 2018 Apr 24. PMID 29691757